CLINICAL TRIAL: NCT00652132
Title: A Multi-centre Open-label Randomised Phase III Trial of the Efficacy of Sodium Thiosulphate in Reducing Ototoxicity in Patients Receiving Cisplatin Chemotherapy for Standard Risk Hepatoblastoma
Brief Title: Cisplatin With or Without Sodium Thiosulfate in Treating Young Patients With Stage I, II, or III Childhood Liver Cancer
Acronym: SIOPEL6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Childhood Liver Tumours Strategy Group - SIOPEL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_09-205; CDR0000590649 (Other: PDQ (Physician Data Query)); 2007-002402-21 (EudraCT Number); SIOP-CCLG-LT-2007-03 (Other: CCLG - previous Sponsor)
Record Dates: First submitted 2008-04-02; First posted 2008-04-03 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Liver Cancer; Ototoxicity
Keywords: ototoxicity; childhood hepatoblastoma; stage I childhood liver cancer; stage II childhood liver cancer; stage III childhood liver cancer
MeSH Terms: conditions — Liver Neoplasms; Ototoxicity; Hepatoblastoma | interventions — Cisplatin; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cisplatin) (Active Comparator): Neoadjuvant and adjuvant cisplatin: patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 2 weeks for 4 courses. Patients with progressive disease after course 4 are taken off study. Patients without evidence of disease progression proceed to surgery. Beginning within 3 weeks after surgery, patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin
- Arm II (cisplatin + STS) (Experimental): Neoadjuvant and adjuvant cisplatin and sodium thiosulphate (STS): patients receive cisplatin IV over 6 hours and sodium thiosulphate IV over 15 minutes (beginning 6 hours after completion of cisplatin) on day 1. Treatment repeats every 2 weeks for 4 courses. Patients with progressive disease after course 4 are taken off study. Patients without evidence of disease progression proceed to surgery. Beginning within 3 weeks after surgery, patients receive cisplatin IV over 6 hours and sodium thiosulphate IV over 15 minutes (as in neoadjuvant therapy) on day 1. Treatment repeats every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: sodium thiosulfate

INTERVENTIONS:
Drug: cisplatin
Drug: sodium thiosulfate
  Arms: Arm II (cisplatin + STS)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as sodium thiosulfate, may protect normal cells from the side effects of chemotherapy. It is not yet known whether giving sodium thiosulfate is effective in reducing hearing damage caused by cisplatin in treating young patients with liver cancer.

PURPOSE: This randomized phase III trial is studying how well sodium thiosulfate works to decrease hearing loss caused by cisplatin in treating young patients with stage I, stage II, or stage III childhood liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy of sodium thiosulfate (STS) to reduce the hearing impairment caused by cisplatin chemotherapy.

Secondary

* To carefully monitor any potential impact of STS on response to cisplatin and survival.
* To assess the short- and long-term tolerability of the combination of STS and cisplatin
* To prospectively evaluate and validate biological, radiological and pathological features of standard-risk hepatoblastoma for future risk adapted management
* To investigate the effect of STS on the formation of cisplatin-DNA adducts.
* To prospectively collect patient DNA specifically for the analysis of possible genetic factors that may contribute to the development of treatment-related ototoxicity and nephrotoxicity

OUTLINE: This is a multicenter study. Patients are stratified according to country, median age (< 15 months vs ≥ 15 months), and PRETEXT tumor classification (I vs II vs III). Patients are randomized to 1 of 2 treatment arms.

* Arm I (Neoadjuvant and adjuvant cisplatin): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 2 weeks for 4 courses. Patients with progressive disease after course 4 are taken off study. Patients without evidence of disease progression proceed to surgery. Beginning within 3 weeks after surgery, patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (Neoadjuvant and adjuvant cisplatin and sodium thiosulphate): Patients receive cisplatin IV over 6 hours and sodium thiosulphate IV over 15 minutes (beginning 6 hours after completion of cisplatin) on day 1. Treatment repeats every 2 weeks for 4 courses. Patients with progressive disease after course 4 are taken off study. Patients without evidence of disease progression proceed to surgery. Beginning within 3 weeks after surgery, patients receive cisplatin IV over 6 hours and sodium thiosulphate IV over 15 minutes (as in neoadjuvant therapy) on day 1. Treatment repeats every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection and tumor biopsies periodically for biological and pharmacological studies consisting of biomarker analysis, gene expression profiling, IHC, proteomic analysis, and gene rearrangement analysis. Patients undergo auditory evaluations at baseline, and at the completion of study treatment or at an age of at least 3.5 years to measure ototoxicity and hearing impairment.

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Histologically confirmed newly diagnosed hepatoblastoma

* Standard risk hepatoblastoma (Pretext I,II,III)
* Age ≤ 18 years and > 1 month
* Written informed consent and national/local ethics committee and regulatory approval
* Centre/country willing and able to organise audiometry at the minimum required quality standard and to provide the contact details of the Consultant Audiologist or Ear Nose and Throat Surgeon who will take the responsibility for seeing that this is done
* Ability to comply with requirements for submission of material for central review
* For females of child-bearing potential, a negative pregnancy test prior to study treatment is required.
* Any patient who is of reproductive age should agree to use adequate contraception for the duration of the trial.

Exclusion:

High risk hepatoblastoma

* Hepatocellular carcinoma
* Treatment starting more than 15 days from written biopsy report
* Abnormal renal function
* Any previous chemotherapy
* Recurrent disease
* Previous hypersensitivity to STS
* Patient unable to follow the protocol for any reason

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2007-12-15 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of Brock grade ≥ 1 hearing loss | End of trial treatment or at an age of 3.5 years, whichever is later
  To investigate if the administration of sodium thiosulfate simultaneously with the administration of Cisplatin significantly reduces the hearing impairment

SECONDARY OUTCOMES:
Response to preoperative chemotherapy | Following completion of preoperative chemotherapy
  Defined as:
  Complete response (CR):
  no evidence of disease and normal serum AFP value (for age).
  Partial response (PR):
  any tumour volume shrinkage associated with a decreasing serum AFP value, > 1 log below the original measurement.
  Stable disease (SD):
  no tumour volume change and no change, or < 1 log fall of the serum AFP concentration.
  Progressive disease (PD):
  unequivocal increase in 1 or more dimensions and/or any unequivocal increase of the serum AFP concentration (three successive 1-2 weekly determinations) even without clinical (physical and/or radiological) evidence of tumour re-growth.
Complete resection | Within 2 weeks after surgery.
  Total macroscopic removal of the tumour as reported by the surgeon and pathologist. In case of any doubt the lack of residual tumour must be confirmed with imaging studies performed
Complete remission | End of trial treatment
  Lack of evidence of residual disease and normal (for age) alpha-foetal protein (AFP). To establish a complete remission all of the following requirements must be fulfilled:
  * No evidence of tumour intra-abdominally: negative abdominal (including hepatic) ultrasound or CT scan or Magnetic resonance imaging
  * No evidence of metastases: clear chest X-ray (PA and lateral) for non-metastatic patients. (Normal lung CT scan for patients with lung metastasis at diagnosis, who are high-risk by definition and not treated according to SIOPEL 6).
  * Serum AFP level either normal or compatible with age for at least 4 weeks after normalisation.
Event-free survival (EFS) | Until first event or up to 5 years
  Calculated from the time of randomisation to the first of the following events: progression, relapse, secondary primary malignancy or death.
Overall survival (OS) | Until event or up to 5 years
  Calculated from the time of randomisation to death.
Toxicity as graded by CTCAE v 3.0 | 30 days post treatment
  Adverse drug reactions are defined as adverse events, which are possibly, probably or definitely related to the trial treatment. They will be assessed according to NCI CTCAE v 3.0.
Long-term renal clearance | Until event or up to 5 years
  By clearance method either EDTA, iohexol or inulin.
Feasibility of central audiology review | End of trial treatment or at an age of 3.5 years, whichever is later
  The feasibility of central review

CONTACTS AND LOCATIONS:
Overall Officials: Milind D. Ronghe, MD, Principal Investigator — Royal Hospital for Sick Children
Locations (16):
- United Kingdom (16):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Childre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Royal Marsden - London, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Queen's Medical Centre, Nottingham, England
  - Sheffield Hallam University - City Campus, Sheffield, England
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - The Noah's Ark Children's Hospital for Wales, Cardiff
  - Royal Hospital For Sick Children, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital Trust, Liverpool
  - John Radcliffe Hospital, Oxford
  - Southampton Children's Hospital, Southampton

REFERENCES:
- [Derived] Brock PR, Maibach R, Childs M, Rajput K, Roebuck D, Sullivan MJ, Laithier V, Ronghe M, Dall'Igna P, Hiyama E, Brichard B, Skeen J, Mateos ME, Capra M, Rangaswami AA, Ansari M, Rechnitzer C, Veal GJ, Covezzoli A, Brugieres L, Perilongo G, Czauderna P, Morland B, Neuwelt EA. Sodium Thiosulfate for Protection from Cisplatin-Induced Hearing Loss. N Engl J Med. 2018 Jun 21;378(25):2376-2385. doi: 10.1056/NEJMoa1801109. PMID 29924955